CLINICAL TRIAL: NCT07159152
Title: Effects of Coffee Versus Hibiscus Tea Consumption During Prolonged Sitting on Blood Pressure and Heart Rate
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: Princess Nourah bint Abdulrahman University, Riyadh, Saudi Arabia (Unknown)
Responsible Party: Principal Investigator, Abdullah Bandar Alansare, Assistant Professor of Exercise Physiology, King Saud University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: No. E-25-9503
Record Dates: First submitted 2025-08-23; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
Keywords: hibiscus drink; coffee; prolonged sitting; sedentary behavior; cardiovascular health; vascular function; cardiovascular regulation
MeSH Terms: conditions — Hypertension; Sedentary Behavior | interventions — Coffee

STUDY DESIGN:
Intervention Model Description: A randomized crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coffee plus prolonged sitting protocol (Experimental): all participants in this group follow the coffee protocol
  Interventions: Dietary Supplement: Coffee
- Hibiscus drink plus prolonged sitting protocol (Experimental): all participants in this group follow the hibiscus drink protocol
  Interventions: Dietary Supplement: Hibiscus drink

INTERVENTIONS:
Dietary Supplement: Coffee — Participants will consume 3 cups of Arabica coffee (Guatemalan origin), providing a total of 400 mg of caffeine. Each cup is prepared with 6% coffee grounds per 100 mL of water, brewed at 90°C for 6 minutes using an electric drip coffee maker, yielding 100.8 mg caffeine per 100 mL. Immediately following coffee consumption, participants will engage in uninterrupted sitting for 3 hours. Blood pressure, heart rate, and other study questionnaires will be measured at baseline (before coffee), 1 hour after coffee intake, and hourly during the 3-hour sitting period.
  Arms: Coffee plus prolonged sitting protocol
Dietary Supplement: Hibiscus drink — Participants will consume 3 servings of hibiscus leaves tea per day, each serving containing 1.25 g of dried hibiscus leaves, totaling 3.75 g per session. The tea will be prepared by steeping the leaves in 240 mL of boiling water (100°C) for 10 minutes. Immediately after consuming the hibiscus tea, participants will engage in uninterrupted sitting for 3 hours. Blood pressure, heart rate, and other study questionnaires will be measured at baseline (before tea), 1 hour after tea intake, and hourly during the 3-hour sitting.
  Arms: Hibiscus drink plus prolonged sitting protocol

SUMMARY:
Modern lifestyles often involve long periods of sitting, which can increase the risk of heart problems, obesity, and other health issues. Diet also plays a key role in heart health. Coffee and hibiscus tea are two common beverages, but their effects during prolonged sitting are not well understood.

This study will examine how drinking coffee versus hibiscus tea affects blood pressure, heart rate, and heart rate variability in men and women during extended periods of sitting.

Participants (30 in total: 15 women and 15 men) will take part in a randomized crossover study, meaning each person will try both beverages at different times. Data will be collected using questionnaires, body measurements, and devices to measure heart rate, blood pressure, and heart rate variability.

The goal is to better understand how these drinks influence heart health during sedentary behavior.

DETAILED DESCRIPTION:
Modern lifestyles, shaped by technological advancements and urbanization, have led to a dramatic increase in sedentary behavior, particularly prolonged sitting. Physical inactivity is a major risk factor for cardiovascular diseases (CVDs), obesity, and premature mortality, with women generally being less active than men. Prolonged sitting affects key indicators of cardiovascular health, including blood pressure, heart rate, and heart rate variability (HRV), which reflect autonomic nervous system regulation and overall heart function. Despite the growing concern, research on how sedentary behavior specifically affects women, particularly in Saudi Arabia, remains limited.

Dietary habits also play a critical role in cardiovascular health. Coffee, one of the most widely consumed beverages worldwide, contains caffeine and polyphenols that can both stimulate and protect the cardiovascular system. Moderate coffee consumption may provide benefits such as reduced risk of chronic diseases and lower resting heart rate, while excessive intake can increase blood pressure, particularly in hypertensive individuals. Hibiscus tea, rich in flavonoids and antioxidants like anthocyanins, has been traditionally used as an antihypertensive agent. It has potential therapeutic effects, including lowering blood pressure, improving metabolic health, and protecting against cardiovascular inflammation. However, the acute effects of these beverages during prolonged sitting are not well understood.

This study aims to investigate the effects of coffee versus hibiscus tea on blood pressure, heart rate, and HRV in healthy women during extended periods of sitting. Using a randomized crossover design, participants will consume each beverage at separate times while their cardiovascular responses are monitored. Data will be collected through questionnaires, body composition measurements, and non-invasive devices to track blood pressure and heart rate variability. By comparing the acute effects of coffee and hibiscus tea during sedentary behavior, this study seeks to provide new insights into how common dietary choices may influence cardiovascular function and help guide recommendations for healthier lifestyles in populations at risk of prolonged sitting.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years.
* Normal to elevated blood pressure (systolic <130 mmHg and diastolic <80 mmHg) and normal resting heart rate (60-100 bpm), ensuring selection of healthy adults and minimizing confounding factors.
* Generally healthy, without chronic or acute medical conditions, to reduce external influences on study outcomes.
* Physically inactive, not meeting current physical activity guidelines, as the study targets sedentary individuals.

Exclusion Criteria:

* Known allergy or hypersensitivity to hibiscus or coffee, as participants will consume these beverages during the study.
* Current use of medications that could influence blood pressure, heart rate, or heart rate variability, including antihypertensive, chronotropic, or vasoactive drugs.
* Any medical condition or health issue that may interfere with safe participation or affect study measurements.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure | Blood pressure will be recorded at five standardized time points: prior to consumption of coffee or hibiscus tea, one hour post-consumption, and following one, two, and three hours of prolonged sitting.
  Systolic and diastolic blood pressure will be assessed using an oscillometric blood pressure monitor (Omron HEM 7124 CP, Omron Healthcare, Illinois, USA). Measurements will be conducted in accordance with the guidelines of the American Heart Association (AHA) and the American College of Cardiology (ACC).
Heart Rate | Heart rate measurements will be performed at multiple time points during each visit: prior to beverage consumption, one hour post-consumption, and after one, two, and three hours of prolonged sitting.
  Heart rate will be measured using the Polar V800 system, which consists of a wristwatch and a Bluetooth heart rate sensor. The sensor will be positioned on the participant's chest, just below the pectoral muscles. Participants will remain seated quietly for 10 minutes while continuous heart rate data are recorded according to the manufacturer's instructions.
  The clearest five-minute segment of the 10-minute recording will be analyzed using Kubios HRV Premium software to assess heart rate (beat/minute)
NN Intervals | NN Intervals measurements will be performed at multiple time points during each visit: prior to beverage consumption, one hour post-consumption, and after one, two, and three hours of prolonged sitting.
  NN Intervals will be measured using the Polar V800 system, which consists of a wristwatch and a Bluetooth heart rate sensor. The sensor will be positioned on the participant's chest, just below the pectoral muscles. Participants will remain seated quietly for 10 minutes while continuous heart rate data are recorded according to the manufacturer's instructions.
  The clearest five-minute segment of the 10-minute recording will be analyzed using Kubios HRV Premium software to assess NN Intervals (milliseconds)
RMSSD | RMSSD measurements will be performed at multiple time points during each visit: prior to beverage consumption, one hour post-consumption, and after one, two, and three hours of prolonged sitting.
  RMSSD will be measured using the Polar V800 system, which consists of a wristwatch and a Bluetooth heart rate sensor. The sensor will be positioned on the participant's chest, just below the pectoral muscles. Participants will remain seated quietly for 10 minutes while continuous heart rate data are recorded according to the manufacturer's instructions.
  The clearest five-minute segment of the 10-minute recording will be analyzed using Kubios HRV Premium software to assess RMSSD (milliseconds squared)

OTHER OUTCOMES:
Height | One time at baseline
  Height (cm) will be measured using an electronic stadiometer (Stadium Scale) with participants standing barefoot in an upright position.
  Measurements will be performed under standardized conditions, with participants wearing light clothing and no shoes, to ensure accuracy and consistency.
Weight | One time at baseline
  Body weight (kg) will be recorded using a calibrated digital scale (Seca).
  Measurements will be performed under standardized conditions, with participants wearing light clothing and no shoes, to ensure accuracy and consistency.
Body Mass Index | One time at baseline
  Body mass index (BMI) (kg/m2) will be calculated based on height and weight.
  Measurements will be performed under standardized conditions, with participants wearing light clothing and no shoes, to ensure accuracy and consistency.
Body Fat Percentage | One time at baseline
  Body fat percentage (%) will be assessed using a bioelectrical impedance analysis device (Tanita MC-980, Japan).
  Measurements will be performed under standardized conditions, with participants wearing light clothing and no shoes, to ensure accuracy and consistency.
Demographic and Personal Information | One time at baseline
  Participant demographic and personal data will be collected using a general information form, which includes age and medical history
Physical activity status | One time at baseline
  Participants will complete the short form of the International Physical Activity Questionnaire (IPAQ). They will report the number of days per week and the average minutes per day they engaged in moderate or vigorous physical activity during the past seven days. These responses will be used to calculate the total minutes per week of moderate-to-vigorous physical activity (MVPA). Participants will then be classified into two groups: those who meet the recommended guideline of at least 150 minutes of MVPA per week, and those who do not meet this guideline (<150 minutes per week).

CONTACTS AND LOCATIONS:
Overall Officials: Hadeel M Almalki, BSc, Principal Investigator — Princess Nourah Bint Abdulrahman University
Locations (1):
- Princess Nourah University Lifestyle Center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside the research team due to restrictions in the informed consent provided by participants

REFERENCES:
- [Result] Abdelmonem M, Ebada MA, Diab S, Ahmed MM, Zaazouee MS, Essa TM, ElBaz ZS, Ghaith HS, Abdella WS, Ebada M, Negida A. Efficacy of Hibiscus sabdariffa on Reducing Blood Pressure in Patients With Mild-to-Moderate Hypertension: A Systematic Review and Meta-Analysis of Published Randomized Controlled Trials. J Cardiovasc Pharmacol. 2022 Jan 1;79(1):e64-e74. doi: 10.1097/FJC.0000000000001161. PMID 34694241
- [Result] Ellis LR, Zulfiqar S, Holmes M, Marshall L, Dye L, Boesch C. A systematic review and meta-analysis of the effects of Hibiscus sabdariffa on blood pressure and cardiometabolic markers. Nutr Rev. 2022 May 9;80(6):1723-1737. doi: 10.1093/nutrit/nuab104. PMID 34927694
- [Result] Da-Costa-Rocha I, Bonnlaender B, Sievers H, Pischel I, Heinrich M. Hibiscus sabdariffa L. - a phytochemical and pharmacological review. Food Chem. 2014 Dec 15;165:424-43. doi: 10.1016/j.foodchem.2014.05.002. Epub 2014 May 27. PMID 25038696
- [Result] Sindi HA, Marshall LJ, Morgan MR. Comparative chemical and biochemical analysis of extracts of Hibiscus sabdariffa. Food Chem. 2014 Dec 1;164:23-9. doi: 10.1016/j.foodchem.2014.04.097. Epub 2014 May 6. PMID 24996300
- [Result] Nohara-Shitama Y, Adachi H, Enomoto M, Fukami A, Nakamura S, Kono S, Morikawa N, Sakaue A, Hamamura H, Toyomasu K, Fukumoto Y. Habitual coffee intake reduces all-cause mortality by decreasing heart rate. Heart Vessels. 2019 Nov;34(11):1823-1829. doi: 10.1007/s00380-019-01422-0. Epub 2019 May 6. PMID 31062117
- [Result] Nurminen ML, Niittynen L, Korpela R, Vapaatalo H. Coffee, caffeine and blood pressure: a critical review. Eur J Clin Nutr. 1999 Nov;53(11):831-9. doi: 10.1038/sj.ejcn.1600899. PMID 10556993
- [Result] Alfawaz HA, Khan N, Yakout SM, Khattak MNK, Alsaikhan AA, Almousa AA, Alsuwailem TA, Almjlad TM, Alamri NA, Alshammari SG, Al-Daghri NM. Prevalence, Predictors, and Awareness of Coffee Consumption and Its Trend among Saudi Female Students. Int J Environ Res Public Health. 2020 Sep 25;17(19):7020. doi: 10.3390/ijerph17197020. PMID 32992846
- [Result] Rao NZ, Fuller M, Grim MD. Physiochemical Characteristics of Hot and Cold Brew Coffee Chemistry: The Effects of Roast Level and Brewing Temperature on Compound Extraction. Foods. 2020 Jul 9;9(7):902. doi: 10.3390/foods9070902. PMID 32659894
- [Result] Hecimovic I, Belscak-Cvitanovic A, Horzic D, Komes D. Comparative study of polyphenols and caffeine in different coffee varieties affected by the degree of roasting. Food Chem. 2011 Dec 1;129(3):991-1000. doi: 10.1016/j.foodchem.2011.05.059. Epub 2011 May 15. PMID 25212328
- [Result] Paterson C, Fryer S, Zieff G, Stone K, Credeur DP, Barone Gibbs B, Padilla J, Parker JK, Stoner L. The Effects of Acute Exposure to Prolonged Sitting, With and Without Interruption, on Vascular Function Among Adults: A Meta-analysis. Sports Med. 2020 Nov;50(11):1929-1942. doi: 10.1007/s40279-020-01325-5. PMID 32757163
- [Result] Taylor FC, Pinto AJ, Maniar N, Dunstan DW, Green DJ. The Acute Effects of Prolonged Uninterrupted Sitting on Vascular Function: A Systematic Review and Meta-analysis. Med Sci Sports Exerc. 2022 Jan 1;54(1):67-76. doi: 10.1249/MSS.0000000000002763. PMID 34334722
- [Result] Vranish JR, Young BE, Kaur J, Patik JC, Padilla J, Fadel PJ. Influence of sex on microvascular and macrovascular responses to prolonged sitting. Am J Physiol Heart Circ Physiol. 2017 Apr 1;312(4):H800-H805. doi: 10.1152/ajpheart.00823.2016. Epub 2017 Jan 27. PMID 28130340
- [Result] Dempsey PC, Larsen RN, Dunstan DW, Owen N, Kingwell BA. Sitting Less and Moving More: Implications for Hypertension. Hypertension. 2018 Nov;72(5):1037-1046. doi: 10.1161/HYPERTENSIONAHA.118.11190. No abstract available. PMID 30354827
- [Result] Adams NT, Paterson C, Poles J, Higgins S, Stoner L. The Effect of Sitting Duration on Peripheral Blood Pressure Responses to Prolonged Sitting, With and Without Interruption: A Systematic Review and Meta-Analysis. Sports Med. 2024 Jan;54(1):169-183. doi: 10.1007/s40279-023-01915-z. Epub 2023 Sep 8. PMID 37682412

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT07159152/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT07159152/ICF_001.pdf